CLINICAL TRIAL: NCT04016207
Title: Non-interventional Trial to Investigate the Change of Psychopathological Markers of Affective Dysregulation (AD) in Children With Attention Deficit Hyperactivity Disorder (ADHD) Treated by Guanfacin, a Pilot Trial
Brief Title: Affective Dysregulation (AD) in Children With ADHD Treated by Guanfacin
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Prof. Dr. Veit Roessner and PD Dr. Robert Waltereit jointly lead and conduct the study (Unknown)
Responsible Party: Principal Investigator, PD Dr. med. Robert Waltereit, Consultant, Technische Universität Dresden
Other Study IDs: IIR-DEU-002258
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Affective Dysregulation
MeSH Terms: interventions — Guanfacine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Guanfacin regular treatment
  Interventions: Drug: Guanfacine

INTERVENTIONS:
Drug: Guanfacine — regular treatment

SUMMARY:
Early onset, high prevalence and persistence, as well as developmental comorbidity make affective dysregulation (AD) in childhood one of the most psychosocially impairing and cost-intensive mental conditions. Despite continuous research, there is still a substantial need for optimization of individual treatment strategies in order to improve outcomes and to reduce subjective and economic burden. Here we want to study the change of psychopathological markers of affective dysregulation (AD) treatment of affective dysregulation (AD) in children with Attention Deficit Hyperactivity Disorder (ADHD) treated by Guanfacine. These children did not respond to methylphenidate treatment. The results will allow the generation of a hypothesis for a randomized clinical trial to investigate the efficacy and safety of Guanfacine for the treatment of AD in children.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients (aged 6 to 17 years)
* clinical diagnosis of ADHD (F90.0) or comorbid ADHD and Oppositional defiant disorder (ODD) (F90.1)
* patients with ADHD who did not respond to stimulants
* DADYS is an instrument to assess AD and has a domain for disruptive behaviors. Inclusion criterion for the study is a score of at least moderate (middle) severity in the DADYS parents version this domain
* IQ must be at least 70
* Patients receiving or intended to receive Guanfacin
* Written informed consent by the custodian and the children

Exclusion Criteria:

* unipolar depression, bipolar disorder, schizophrenia or any other psychotic disorder
* current substance abuse

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with the diagnosis of ADHD, Age 6-17 years
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
DADYS-EF (Diagnostikum für Affektive Dysregulation, Eltern-Fragebogen) | 9 weeks
  The DADYS is a German instrument to assess affective dysregulation. The Eltern-Fragebogen is the parents' version of the rating scale.

SECONDARY OUTCOMES:
DADYS-KF (Diagnostikum für Affektive Dysregulation, Kinder-Fragebogen) | 9 weeks
  The DADYS is a German instrument to assess affective dysregulation. The Kinder-Fragebogen is the childrens' version of the rating scale.
Conners3L | 9 weeks
  The Conners 3rd Edition™ (Conners 3®) is a thorough assessment of attention-deficit/hyperactivity disorder (ADHD) and its most common comorbid problems and disorders in children and adolescents aged 6 to 18 years. It is a multi-informant assessment that takes into account home, social, and school settings, with rating forms for parents, teachers, and youth.

CONTACTS AND LOCATIONS:
Overall Officials: Veit Roessner, MD, Study Director — Technical University Dresden, Child and Adolescent Psychiatry

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Waltereit J, Uhlmann A, Tarassidis C, Preuss U, Roessner V, Waltereit R. Treatment of affective dysregulation in ADHD with guanfacine: study protocol. Front Child Adolesc Psychiatry. 2025 Mar 28;4:1547672. doi: 10.3389/frcha.2025.1547672. eCollection 2025. PMID 40226438